CLINICAL TRIAL: NCT05576363
Title: Food Security Status and Its Association With Maternal Nutrition and Birth Outcomes Among Low Income Mothers in Kota Kinabalu, Sabah
Brief Title: Food Security and Maternal Nutrition Status
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Universiti Malaysia Sabah (Other)
Responsible Party: Principal Investigator, Dr. Bibi Nabihah Abdul Hakim, Principal Investigator, Universiti Malaysia Sabah
Other Study IDs: UMalaysiaSabah
Record Dates: First submitted 2022-09-08; First posted 2022-10-12 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Pregnancy Related
Keywords: Food security, Pregnancy, Nutritional status, Infant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Maternal: Second trimester

SUMMARY:
Food insecurity has been climbing slowly for several recent years and affects more than 30% of the world population in 2021. Poor households tend to have poor diet quality in accordance to expensive price of food, thus reduce dietary diversity. They frequently consume low-cost foods that are high in energy density but low in micronutrient content, diets that are poor in fruits, vegetables, milk, and dairy products, and eating habits that are unhealthy. The double burden malnutrition will affect pregnant women who were vulnerable due to increase demand of nutrition during pregnancy and also their infants. Food insecurity has been linked to maternal stress, weight gain, gestational diabetes, low birth weight, birth defects, premature birth, hospitalization of infants aged less than 6 months and cause the long-term consequences for child growth and development. Therefore, this study aimed to examine the level of food security and its association with maternal nutrition and birth outcomes. This prospective cohort study will be conducted among 150 pregnant women (in 2nd trimester) at government health clinic near Kota Kinabalu. The participants will be assessed on sociodemographic data, socio-economic, medical history, anthropometry measurements, food security, dietary intake and stress level at baseline. After 6 months, birth outcomes will be recorded. The expected outcomes will be that there will be high prevalence of food insecurity among pregnant mother. Besides, the food insecure mothers will be associated with poor nutritional status and have negative consequences on birth outcomes (low birth weight and short stature). This study will highlight the level of food insecurity to inform much needed interventions to address important global health challenges of nutrition and could improve the prenatal care.

DETAILED DESCRIPTION:
The burden of food insecurity on maternal nutritional status is understudied. This will underestimate the negative consequences on maternal health and infant. Even though the mechanisms by which food security influences pregnancy outcomes remains unclear, the association between food security and maternal nutritional status warrants further exploration. This prospective study will provide a novel data with the potential to inform that there is much needed interventions to address these important global health challenges.

Therefore, the proposed study is to advocate the evidence-based and obtain a more comprehensive picture of the impact of food security on maternal nutrition and birth outcomes. The prevalence of food security and the risks of malnutrition among maternal and neonates will be explored further. Based on the potential for food insecurity and the effects on maternal health and birth outcomes, screening in primary care settings may help providers to identify the needs and to address the issues through referrals to additional resources.

This is a prospective cohort study design will be conducted among pregnant women in the second trimester at government health clinic located at Kota Kinabalu, Sabah.

Study location:

Randomly selected health clinic near Kota Kinabalu Sabah.

Duration of study:

The study will be conducted from September 2022 to September 2024. The data collection will be held in health clinic in between February 2023 and February 2024.

Tools:

1. Sociodemographic, Socio-economic, medical history, anthropometry measurements of maternal and infant
2. Radimer/Cornell Item Assessment of food security status of pregnant mother.
3. 24-hour dietary recall (3 days) Nutritional assessment were recorded to assess the adequacy of nutrient intake by pregnant women.
4. Knowledge, Attitude and Practice (KAP) of maternal nutrition Nutritional knowledge among pregnant women may reflect the quality of food intake and also healthy food choices.
5. Perceive Stress Scale (PSS-10) questionnaire

ELIGIBILITY:
Inclusion Criteria:

* In second trimester (13-27 weeks of pregnancy)
* B40 income group (<RM3490) as categorized for population in Kota Kinabalu, Sabah
* Aged 18-39 years old
* Malaysian
* Have no/controlled medical illness

Exclusion Criteria:

* Multiple pregnancy
* Uncontrolled medical illness
* Have pregnancy complications

Ages: 18 Years to 39 Years | Sex: Female
Age Groups: Adult
Study Population: Pregnant mother at second trimester
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-07-28 (Estimated); Primary Completion 2023-07-28 (Estimated); Study Completion 2024-08-15 (Estimated)

PRIMARY OUTCOMES:
Level of food security level and nutritional status of pregnant mothers in Kota Kinabalu, Sabah. | January 2023- June 2023
  Assessment food security by using Radimer Cornell Food Insecurity Questionnaire and 3 days diet recall for nutritional status

SECONDARY OUTCOMES:
Association between level of food security and nutritional status status. | January 2023- June 2023
  Assess the association of food security on anthropometry and dietary data using correlation

OTHER OUTCOMES:
Association between maternal nutritional status and birth outcomes outcomes. | January 2024- April 2024
  Assess association between maternal nutritional status and birth outcome (anthropometry of infant)

CONTACTS AND LOCATIONS:
Overall Officials: DR. BIBI NABIHAH ABDUL HAKIM, PHD, Principal Investigator — Universiti Malaysia Sabah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1. Life Science Research Office Expert Panel, National Research Council. The federation of American societies for experimental biology. In: Wunderlich GS, Norwood JL, editors. Food insecurity and hunger in the United States: an assessment of the measure. Washington, DC: National Academies Press; 1990. pp. 13-54.